CLINICAL TRIAL: NCT02425254
Title: Preemptive Paracetamol for Postoperative Pain: a Randomised, Double-blind, Two Way Crossover Trial
Brief Title: Preemptive Paracetamol for Postoperative Pain
Acronym: PPPP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15029
Record Dates: First submitted 2015-04-09; First posted 2015-04-23 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Pain; Surgical Wound
MeSH Terms: conditions — Pain; Surgical Wound

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Preemptive paracetamol (Experimental): 1000mg intravenous paracetamol given ≥15 minutes before surgical incision and intravenous saline 15 minutes before the end of surgery
  Interventions: Drug: Intravenous paracetamol; Drug: Intravenous saline 0.9%
- Postincision paracetamol (Active Comparator): Intravenous saline ≥15 minutes before surgical incision and 1000mg intravenous paracetamol given 15 minutes before the end of surgery
  Interventions: Drug: Intravenous paracetamol; Drug: Intravenous saline 0.9%

INTERVENTIONS:
Drug: Intravenous paracetamol — 1000mg intravenous solution for infusion
Drug: Intravenous saline 0.9% — 0.9% sodium chloride in order to ensure double-blinding

SUMMARY:
The purpose of this study is to test whether a dose of paracetamol given before surgical incision is more effective at reducing postoperative pain and analgesic consumption in cervical spine surgery versus a dose given at the end of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 years old
* Patients listed for non-malignant cervical spinal surgery
* General anaesthesia
* Capacity to give informed consent
* Ability to use PCA device and pain score scale
* ASA I, II and III
* >50kg in weight

Exclusion Criteria:

* Allergy or sensitivity to paracetamol, proparacetamol or morphine
* Liver disease
* Renal disease (creatinine clearance <30ml/min)
* Bleeding disorder
* Chronic alcoholism
* Chronic malnutrition
* Dehydration
* G6PD deficiency
* Hypernatraemia (Na >150)
* Hypokalaemia (K <3.5) and hyperchloraemia
* Pregnancy or breast-feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Morphine consumption | 24 hours postoperatively
  Measured from PCA machine

SECONDARY OUTCOMES:
Time to first analgesic request | 24 hours
  In minutes
Nausea and vomiting | 24 hours
  Incidence of nausea or vomiting 24 hours postoperatively
Pruritus | 24 hours
  Incidence of pruritus 24 hours postoperatively
Sedation | 24 hours
  Incidence of sedation 24 hours postoperatively
Urinary retention | 24 hours
  Incidence of urinary retention 24 hours postoperatively
Allergic reaction | 24 hours
  Incidence of allergic reaction (defined as diagnosed by clinician 24 hours postoperatively)
Pain score | 1 hour
  Numeric rating scale (NRS)
Pain score | 2 hours
  Numeric rating scale (NRS)
Pain score | 6 hours
  Numeric rating scale (NRS)
Pain score | 12 hours
  Numeric rating scale (NRS)
Pain score | 24 hours
  Numeric rating scale (NRS)

CONTACTS AND LOCATIONS:
Overall Officials: John Williams, Principal Investigator — University of Nottiongham